CLINICAL TRIAL: NCT01339156
Title: Randomized, Double-blind, Placebo-controlled Phase I-Ib Study of P3914 to Evaluate the Safety, Tolerability, Food Effect & Pharmacokinetics in Healthy Male Subjects and Efficacy & Safety of P3914 in Patients With Acute Dental Pain
Brief Title: Study of P3914 to Evaluate the Safety, Tolerability, Food Effect & Pharmacokinetics in Healthy Male Subjects and Efficacy & Safety of P3914 in Patients With Acute Dental Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P3914/48/10
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Acute Dental Pain
Keywords: Safety; Tolerability; Food Effect; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- P3914 (Experimental)
  Interventions: Drug: P3914
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P3914 — Part A:
  The subjects will be fasted overnight for at least 10 hrs.The drug will be administered orally to each subject in sitting posture.
  Part B:
  Dosing will start on Day 1. Each subject will receive the investigational product under fasting conditions for 14 days (Days 1 to 14).
  The investigational product will be administered orally to each subject with 240 mL of water.
  Part C:
  Dosing will take place on Day 1 of each study period. Each subject will receive a single oral dose.
  For administration of P3914 tablets subjects will be required to fast for 10 hrs prior to dosing.
  Part D:
  Patients will be fasted for at least 4-6 hrs. The investigational product will be administered orally to each subject in sitting posture on day 1 within 6 hrs of first administration of anesthesia (day of dental surgery).
  Arms: P3914
Drug: Placebo — Part A:
  The subjects will be fasted overnight for at least 10 hrs. The investigational product (allocated as per the randomisation schedule) will be administered orally to each subject in sitting posture.
  Part B:
  Dosing will start on Day 1. It is planned that each subject will receive the investigational product under fasting conditions for 14 days (Days 1 to 14).
  The investigational product (allocated as per the randomisation schedule) will be administered orally to each subject with 240 mL of water.
  Part D:
  Patients will be fasted for at least 4-6 hrs. The investigational product (allocated as per the randomisation schedule) will be administered orally to each subject in sitting posture on day 1 within 6 hrs of first administration of anesthesia (day of dental surgery).
  Arms: Placebo

SUMMARY:
P3914 a pro-drug of Naproxen, characterized by naproxen (COX inhibiting moiety) linked to a NO moiety is intended for the treatment of pain and inflammation. The rationale behind development of P3914 is to maintain the analgesic, antipyretic and anti-inflammatory activity of naproxen and enhance GI safety by virtue of release of NO besides with no major effect on blood pressure on long-term administration.

ELIGIBILITY:
Inclusion Criteria:

* for Part A, Part B and Part C

  1. Male subjects aged between 18 and 45 years (including both) with Body Mass Index between 18 to 25 kg/m2 (including both).
  2. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable normal range.
  3. Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
  4. Subjects having clinically acceptable X-Ray chest (P/A view).
  5. Subjects having clinically acceptable endoscopy.
  6. Have a negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
  7. Have negative alcohol breath test.
  8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Part D:

Patients with acute postoperative dental pain (at least moderate in severity or score of 40 mm on VAS) after removal of an impacted third mandibular molar will be selected for study participation, if they meet the following criteria:

1. Male patients aged between 18 and 60 years (including both).
2. Patients with acute postoperative dental pain (at least moderate in severity or score of 40 mm on Visual Analogue Scale)
3. Patients with otherwise normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable normal range.
4. Patients having clinically acceptable 12-lead electrocardiogram (ECG).
5. Patients having clinically acceptable chest X-Ray (P/A view).
6. Patients having clinically acceptable endoscopy.
7. Have a negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
8. Have negative alcohol breath test.
9. Patients willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

* Part A, Part B and Part C:

  1. Hypersensitivity to NSAIDs or nitrodonating drugs.
  2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
  3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within one month of the study starting.
  4. History or presence of significant gastric and/or duodenal ulceration including the last three months or gastroduodenal bleeding including the last six months prior to the screening visit.
  5. History of peptic ulceration or significant dyspepsia as judged by the investigator.
  6. Endoscopy finding of gastric or duodenal ulcer at baseline. Erosive esophagitis or other endoscopic appearance that constitutes a risk to the subject, if included in the study, as judged by the investigator.
  7. Have positive test for Helicobacter pylori infection.
  8. Orthostatic hypotension with a systolic blood pressure drop of ≥ 25 mm Hg and/or a diastolic blood pressure drop of ≥ 15 mm Hg within 5 minutes of standing when changing from supine to erect position.
  9. A history of renal impairment, or a glomerular filtration rate (GFR) <60 mL/min or, at visit 1, a serum creatinine value >140 mol/L.
  10. Use of aspirin, H2 antagonists, antacids, misoprostol, proton pump inhibitors, sucralfate including two weeks prior to the screening visit.
  11. Subjects currently taking sildenafil, anticoagulants or ticlopidine, nitrates, nitrovasodilating drugs (e.g. nitroglycerin, isosorbide dinitrate, isosorbide mononitrate, glycerin trinitrate), diuretics (in a dose potentially leading to volume depletion).
  12. Use of any prescribed medication during last two weeks or OTC medicinal products (including herbal/traditional medicine preparations) during the last one week prior to initiation of study.
  13. History or presence of significant alcoholism or drug abuse in the past one year.
  14. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
  15. History or presence of smoking or use of other tobacco, pan, gutkha products since last six months.
  16. History or presence of significant asthma, urticaria or other allergic reactions.
  17. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumour.
  18. Difficulty in swallowing solids like tablets or capsules.
  19. History or presence of cancer.
  20. Difficulty with donating blood.
  21. Major illness during three months before screening.
  22. Participation in a drug research study within past three months.
  23. Donation of blood in the past three months before screening.

For Part D:

1. Hypersensitivity to NSAIDs or nitrodonating drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of significant gastric and/or duodenal ulceration including the last three months or gastroduodenal bleeding including the last six months prior to the screening visit.
5. History of peptic ulceration or significant dyspepsia as judged by the investigator.
6. Endoscopy finding of gastric or duodenal ulcer at baseline. Erosive esophagitis or other endoscopic appearance that constitutes a risk to the subject, if included in the study, as judged by the investigator.
7. Have positive test for Helicobacter pylori infection.
8. Orthostatic hypotension with a systolic blood pressure drop of ≥ 25 mm Hg and/or a diastolic blood pressure drop of ≥ 15 mm Hg within 5 minutes of standing when changing from supine to erect position.
9. A history of renal impairment, or a glomerular filtration rate (GFR) <60 mL/min or, at visit 1, a serum creatinine value >140 mol/L.
10. Use of aspirin, H2 antagonists, antacids, misoprostol, proton pump inhibitors, sucralfate including two weeks prior to the screening visit.
11. Patients currently taking sildenafil, anticoagulants or ticlopidine, nitrates, nitrovasodilating drugs (e.g. nitroglycerin, isosorbide dinitrate, isosorbide mononitrate, glycerin trinitrate), diuretics (in a dose potentially leading to volume depletion).
12. Use of analgesics in the 48 hrs preceding the day of dental surgery except use of acetaminophen until midnight on the day before surgery.
13. Patients with oral surgery in the 30 days before the pre-study visit.
14. Use of any prescribed medication during last two weeks or OTC medicinal products (including herbal preparations) during the last one week prior to initiation of study.
15. History or presence of significant alcoholism or drug abuse in the past one year.
16. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
17. History or presence of smoking or use of other tobacco, pan, gutkha products since last 06 months.
18. History or presence of significant asthma, urticaria or other allergic reactions.
19. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumour.
20. Difficulty in swallowing solids like tablets or capsules.
21. History or presence of cancer.
22. Difficulty with donating blood.
23. Major illness during three months before screening.
24. Participation in a drug research study within past three months.
25. Donation of blood in the past three months before screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Vital signs- systolic and diastolic blood pressure, pulse rate and oral body temperature. | Defined in description
  Vital signs will be measured using DASH 4000. Predose vital signs will be recorded within 30 minutes prior to dosing.
  Part A: pre-dose & at 1,2,3,4,5,6,8,12,16,24,48,72,96 & 120 hrs post dose. Part B:pre-dose on Day 2 to Day 13,predose & at 4 and 12 hrs post-dose on Days 1 &14.Part:C: pre-dose & at 1, 2, 3, 4, 5,6,8,12,24,48,72,96 & 120 hrs postdose.Part D:predose & at 0.5,1,2,4,&8 hrs post dose.

SECONDARY OUTCOMES:
Pain intensity using 100 mm Visual analog scale | immediately before administration of study drug and at 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, and 8.00 hrs post-dose, and immediately before administration of rescue analgesia (if any).
  This assessment will be carried out in Part D of the study.
Pharmacokinetic assessment for Part A | within 15 min prior to dosing. Post-dose blood samples will be drawn at 0.25, 0.50, 1, 2, 3, 3.50, 4, 4.50, 5, 5.50, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96 & 120 hrs following drug administration.
  The concentration time data generated for P3914, naproxen and nitrate/nitrite levels will be used to calculate the following pharmacokinetic parameters as appropriate using non-compartmental analysis tool Tmax, Cmax, AUC0-t, AUC0-inf, AUC0-24h, % AUC Extrapolated, T1/2, kel, CL, Vz.
Pharmacokinetic assessment for Part C | within 15 min prior to dosing. Post-dose samples will be drawn at 0.25, 0.50, 1, 2, 3, 3.50, 4, 4.50, 5, 6, 8, 10, 12, 24, 48, 72, 96 & 120 hrs following drug administration.
  The concentration time data generated for P3914, Naproxen and nitrate/nitrite levels will be used to calculate the following pharmacokinetic parameters as appropriate using non-compartmental analysis tool:• Tmax, Cmax, AUC0-t, AUC0-inf, T1/2, and kel.
Pharmacokinetic assessment for Part B | within 15 min prior to dosing on Day 1, 6, 9, 13&14. Post-dose blood samples at 0.25, 0.50, 1, 2, 3, 3.50, 4, 4.50, 5, 5.50, 6, 8, 10, 12, 16& 24 hrs following drug administration on Day 1 & Day 14 and 48 hrs post-dose on Day 16
  The concentration time data generated for P3914, Naproxen and and nitrate/nitrite levels will be used to calculate the following pharmacokinetic parameters (as appropriate) using non-compartmental analysis tool:
  Tmax, Cmax, AUC0-t, AUC0-inf, AUC0-24h, T1/2, kel, CL, Vz for Day 1 AND Cmax,ss, AUC0-τ,ss, Cmin,ss, Tmax,ss, Cavg,ss Swing, Percent Fluctuation, t1/2 and Kel for Day 14.
Pharmacokinetic assessment for Part D | within 15 min prior to dosing. Post-dose blood samples of at 0.50, 1, 2, 3, 3.50, 4, 4.50, 5, 5.50, 6 and 8 hrs following drug administration
  The concentration time data generated for P3914, Naproxen and nitrate/nitrite levels will be used to calculate the following pharmacokinetic parameters as appropriate using non-compartmental analysis tool:Tmax, Cmax, AUC0-t, AUC0-inf, T1/2, and kel.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dharmesh Domadia, Principal Investigator — Veeda Clinical research private limited